CLINICAL TRIAL: NCT04826952
Title: Malignant Testicular Tumors in Children: A Single Institution's 12-year Experience
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20201912B0
Record Dates: First submitted 2021-03-28; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Overall Survival Rates
Keywords: Testicular tumor, children, histology, orchiectomy, inguinal approach
MeSH Terms: conditions — Testicular Neoplasms | interventions — Orchiectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Orchiectomy — Childhood testicular tumors deserve special diagnostic attention from the therapeutic point of view. A testicular tumor should be considered malignant until proven otherwise. In cases with suspicion of testicular tumors, the inguinal approach is preferred to the scrotal approach for scrotal violation.

SUMMARY:
Background and Objectives. Testicular neoplasms are not commonly found in children, a formidable threat if treated inappropriately. However, there is no consensus concerning their management. The study aimed to present a holistic picture of the integrated treatment of malignant testicular tumors based on our 12 years' experience.

Patients and Methods. This institutional-based retrospective cohort study evaluated clinical presentation, histopathologic diagnosis, treatment, and outcome in 42 boys with malignant neoplasm of testis treated between 2006 and 2019.

DETAILED DESCRIPTION:
Study Design. We retrospectively investigated the outcomes of 42 boys aged 0-19 years presenting with testicular masses. Excluding patients with incomplete records, they were treated at a tertiary referral center between May 2006 and November 2019, which were reviewed and retrospectively analyzed based on their age at the time of admission, presenting complaints, clinical and radiological findings, tumor markers, management, and follow-up. Pathology was centrally reviewed (C.H.) in patients with a tissue biopsy, but confirmation by a central review was not required before enrollment. This retrospective study was unanimously approved by the institutional review board of Chang Gung Memorial Hospital. Their parents or legal guardians provided written informed consent through an opt-out method on our hospital website following the ethical principles for medical research involving human subjects in Taiwan.

Data Collection. The evaluation included age at presentation, medical history, clinical characteristics, diagnostic procedures, treatment methods, histopathologic findings, and outcomes for every patient. All patients received the examinations of color Doppler ultrasonography of the testis and the abdomen, plain x-ray of the thorax, and serum α-fetoprotein (AFP) levels before operations. The AFP measurement is usually very high in newborns and does not decrease to normal adult levels until 8 months. Thus, the AFP levels of infants were evaluated according to reference ranges [4,5].

Surgical Technique All 42 tumors were treated surgically. We explored the groin through an inguinal incision. The testicle is gently grasped and exteriorized, and the spermatic cord and vessels within the tunica vaginalis are clamped. The resected tumor mass was sent for frozen section examination (FSE). Testis-sparing surgery was considered in patients with non-germ cell tumors. If the tumor had replaced the entire testis, a radical orchiectomy was taken. All tumors received histologic analysis. The optimal follow-up protocol included regular control visits with the physical examination, AFP measurements, and testicular sonography. Adjuvant chemotherapy was administered, depending on histopathology and TNM criteria for tumor classification. If non-germ cell tumors were assessed accurately on FSE, testis-sparing surgery could be considered an alternative treatment modality.

ELIGIBILITY:
Inclusion Criteria:

* aged 0-19 years presenting with malignant testicular masses

Exclusion Criteria:

* patients with incomplete records

Ages: 0 Years to 19 Years | Sex: Male
Age Groups: Child, Adult
Gender Based: Yes — We retrospectively investigated the outcomes of 42 boys aged 0-19 years presenting with testicular masses.
Study Population: The evaluation included age at presentation, medical history, clinical characteristics, diagnostic procedures, treatment methods, histopathologic findings, and outcomes for every patient. All patients received the examinations of color Doppler ultrasonography of the testis and the abdomen, plain x-ray of the thorax, and serum α-fetoprotein (AFP) levels before operations. The AFP measurement is usually very high in newborns and does not decrease to normal adult levels until 8 months. Thus, the AFP levels of infants were evaluated according to reference ranges.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
The 1- and 5-year overall survival rates | between May 2006 and November 2019
  Malignant testicular tumors in children:

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Other, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided